CLINICAL TRIAL: NCT02032732
Title: Utilization of Leukocyte Esterase in the Diagnosis of Pediatric Joint Infections
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator resigned from institution
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Other Study IDs: 13-106
Record Dates: First submitted 2013-12-20; First posted 2014-01-10 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Joint Infection; Septic Arthritis
MeSH Terms: conditions — Arthritis, Infectious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- suspected infection: leukocyte esterase test on fluid removed by intra-articular aspiration for suspected infection
  Interventions: Other: leukocyte esterase test
- no suspected infection: leukocyte esterase test on fluid removed by intra-articular aspiration for reason other than suspected infection
  Interventions: Other: leukocyte esterase test

INTERVENTIONS:
Other: leukocyte esterase test — leukocyte esterase test on fluid removed by intra-articular aspiration

SUMMARY:
Pediatric joint infections are a common diagnostic dilemma encountered by treating orthopaedic surgeons. No single test is sensitive or specific enough to stand alone in determining the presence of joint infection.

The purpose of this study is to test the usefulness of a chemical test strip to detect infection in fluid that is removed from a joint (intra-articular aspiration) in pediatric patients. The test strip measures an enzyme called leukocyte esterase, which has been shown to be useful in detecting the presence of infection in fluids from other parts of the body. This study will assess the efficacy of the leukocyte esterase test as a diagnostic tool for evaluating pediatric joint infections. The hypothesis of the study is that a positive leukocyte esterase test identifies a septic joint in pediatric patients undergoing intraoperative joint aspiration.

DETAILED DESCRIPTION:
Pediatric patients requiring an intra-articular joint aspiration for suspected infection or for other reasons will have a leukocyte esterase test performed on fluid removed from the joint. A convenience sample of consecutive patients will be screened according to inclusion/exclusion criteria and enrolled in the study by informed consent. All patients who will be screened for the study will have already been identified as needing an intra-articular joint aspiration in accordance with standard of care. All patients who are enrolled in the study will have the leukocyte esterase test performed on the fluid that is aspirated. Results of the test strip will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* All patients at this facility over the age of 3 months and below the age of 18 years who receive an intra-articular aspiration

Exclusion Criteria:

* Immunocompromised patients
* Renal failure patients
* Patients younger than 3 months old
* Patients 18 years of age or older
* Volume of aspirate is less than 1.5 mL

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patients at a tertiary referral center who will receive an intra-articular aspiration
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
leukocyte esterase level using a leukocyte esterase test strip | at the time of an intraoperative joint aspiration
  A positive leukocyte esterase test strip will be considered an indicator of a septic joint

SECONDARY OUTCOMES:
baseline leukocyte esterase level for pediatric patients using a leukocyte esterase test strip | at the time of intraoperative joint aspiration

CONTACTS AND LOCATIONS:
Overall Officials: Julie Zielinski, M.D., Principal Investigator — UTCOM Chattanooga/Erlanger Health System
Locations (1):
- Children's Orthopaedics, Erlanger Health System, Chattanooga, Tennessee, United States